CLINICAL TRIAL: NCT06690580
Title: The Effect of Motivational Interviews Based on Information, Motivation, Behavioral Skills Model on Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Sevilay Aydın Çelik, MSc, Specialist Nurse, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SBU-SBE-SAC-01
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Breastfeeding Counseling Based on Motivational Interviewing
Keywords: Information, motivation, behavioral skills model; breastfeeding; nursing; motivational interviewing
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- motivational interviews group (Experimental)
  Interventions: Other: Motivational interviewing based on the knowledge motivation behavior skills model
- control group (No Intervention)

INTERVENTIONS:
Other: Motivational interviewing based on the knowledge motivation behavior skills model — Breastfeeding education that includes motivational interviews based on the knowledge motivation behavior skills model
  Arms: motivational interviews group

SUMMARY:
The research is a randomized controlled experimental type and aims to determine the effect of motivational interviews based on the Knowledge, Motivation, Behavioral Skills Model on breastfeeding. The research will be conducted with 90 people (45 experimental, 45 control group) who meet the sample criteria between October 30, 2024 and July 30, 2025. The experimental group will be given breastfeeding training accompanied by motivational interviews, and the control group will not receive any intervention.

DETAILED DESCRIPTION:
Breastfeeding is the healthiest and most effective way for the unique nutrient breast milk to reach the baby. Breastfeeding has many physiological, psychological, social, emotional, societal and economic benefits. Women's inexperience in breastfeeding, the weak value they attribute to breastfeeding, lack of social support systems, and breastfeeding problems they experience can be obstacles to successful breastfeeding. Breastfeeding problems experienced during the lactation process lead to a feeling of exhaustion and inadequacy in the mother and cause mothers to stop breastfeeding. The most common factors that negatively affect breastfeeding are; nipple trauma, breast pain, breast fullness, mastitis, excessive or low breast milk production, difficulty in placing the baby at the breast, breast refusal in the baby, the mother and/or the baby being sick and using medication as a result, fatigue and exhaustion in the mother. Along with these problems, the mother's return to work life is also among the factors that negatively affect breastfeeding. Breastfeeding education and counseling programs are effective in initiating and continuing breastfeeding, solving breastfeeding problems, increasing self-sufficiency, and increasing breastfeeding rates. Nurses, who are important building blocks of the health team, provide support to mothers from the prenatal period to the postnatal period by using their roles as caregivers, decision-makers, patient rights advocates, educators, and consultants. Today, thanks to the development of technology and easy access, traditionally applied trainings have been replaced by trainings provided with newer, modern, visual technologies. These can be listed as peer education, telephone counseling, online and web-based counseling, teach-back, home visits, and model use. Studies have reported that health education programs based on the Information-Motivation-Behavioral Skills Model have a positive effect on individuals' health practices, increase self-sufficiency, and contribute to the development of positive behaviors in individuals. In recent years, motivational interviewing techniques have also been frequently encountered in nursing practices. With the motivational interviewing technique applied during the breastfeeding process, mothers' individual preferences are valued, their indecisiveness is resolved, and their self-sufficiency is supported. In this context, this study aimed to examine the effect of motivational interviews based on the Knowledge, Motivation, Behavioral Skills Model on breastfeeding. The randomized controlled experimental study will be conducted with 90 people (45 experimental, 45 control group) who meet the sampling criteria between October 30, 2024 and July 30, 2025. 4 sessions of motivational interviewing will be applied to the experimental group, and no intervention will be made to the control group. The analysis of the collected data will be done with the SPSS program.

ELIGIBILITY:
Inclusion Criteria:

* Women who speak Turkish,
* Are primigravida,
* Are in their 34th week of pregnancy and above,
* Do not have any chronic disease, diagnosed mental or psychiatric illness,
* Do not have a risky pregnancy,
* Do not have a planned cesarean section were planned to be included in the study.

Exclusion Criteria:

* Women who gave birth by Caesarean section,
* Those who developed complications during birth,
* Those whose baby's birth weight was less than 2500 grams, whose APGAR score was 6 or less at the 5th minute, who were admitted to the neonatal intensive care unit,
* Those who did not attend at least one interview,
* Women who wanted to leave the study were planned to be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women are required to participate.
Enrollment: 90 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy | 10 months
  It is assessed with the Breastfeeding Self-Efficacy Scale-Short Form.The lowest score that can be obtained from the scale is 14, the highest score is 70. Higher scores on the scale indicate higher breastfeeding self-efficacy.

SECONDARY OUTCOMES:
Breastfeeding Motivation | 10 months
  In primiparous women, breastfeeding motivation is evaluated. The "Value Given to Breastfeeding" sub-dimension can receive scores ranging from 13-91 points, the "Self-Efficacy" sub-dimension can receive scores ranging from 7-49 points, and the "Perceived Midwife Support" sub-dimension can receive scores ranging from 4-28 points. The "Expectation of Success" sub-dimension can receive scores ranging from 5-35 points. The evaluation is made by adding the scores obtained in each sub-group in the scale. As the score in the sub-dimension increases, the feature in the sub-dimension and therefore the motivation increases.
Motivational Interviewing Importance and Confidence-Competence Levels | 10 months
  Motivational Interviewing is measured with Importance and Confidence-Competence Scales. scale will evaluate the importance given to breastfeeding, the level of confidence and competence in breastfeeding. The score that can be obtained from the scale varies between 0-10 points. In the importance scale, the individual will be asked the question "How important is breastfeeding to you?" and will be asked to determine the most appropriate score on the scale. A score of 0 means not important at all, and a score of 10 means very important. In the confidence-competence scale, the individual will be asked the question "How confident are you in succeeding in breastfeeding?". They will be asked to give a score between 0-10 to this question. A score of 0 means I do not have confidence at all, and a score of 10 means I have great confidence. The individual will be encouraged to change according to the score they give to the question by discussing the pros and cons.
Breastfeeding Diagnosis | 10 months
  Breastfeeding diagnosis will be made with the LATCH Breastfeeding Diagnostic Measurement Tool. It consists of five evaluation criteria and takes its name from the abbreviation of the first letters of the English equivalents of these criteria. "L; Latch on the breast, A; Audible swallowing, T; Type of the nipple, C; Comfort breast/nipple of the mother and H; Hold/Help position for the baby." Each item is evaluated between 0-2 points. The score that can be obtained from the measurement tool can vary between 0-10, and a high score indicates high breastfeeding success.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University, Istanbul, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No